CLINICAL TRIAL: NCT00983450
Title: The Influences of Watching a Movie Clip of Normal Walking on Measurable Walking Parameters Among Post-brain-stroke Patients as Opposed to the Influences of a Control Movie Clip Showing Backwards Walking
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Zeev Meiner, Hadassah Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0303-09-HMO
Record Dates: First submitted 2009-09-06; First posted 2009-09-24 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2009-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (Experimental): People after a first ischemic or hemorrhagic stroke, up to 60 days following the event.
  Interventions: Other: watching a normal walking clip
- CONTROL (Experimental): People after a first ischemic or hemorrhagic stroke, up to 60 days following the event.
  Interventions: Other: watching walk backward clip

INTERVENTIONS:
Other: watching a normal walking clip — the study group will gain an intervention consisting of 12 therapy sessions, administered for 12 consecutive days (apart of weekends). The intervention will include 6 minutes of watching a movie clip alternately showing a healthy man and a healthy woman at their sixties, walking while being filmed from various angles. Immediately after watching, the subject will perform 6 minutes of walking, under the experimenters supervision, but without his or hers intervention. Immediately following the walking, the whole procedure will be repeated (watching a clip and walking).
  Arms: study group
Other: watching walk backward clip — The control group will undergo 12 treatments of the same nature, but will watch the movie clip shown backwards, so that the people filmed will seem to walk backwards (it was established that watching a reversed action does not activate the MNS system activated by a regular execution of the activity [Celnik et al., 2008]), followed by 6 minutes of walking under the experimenters supervision, then watching the movie again and walking again.
  Arms: CONTROL

SUMMARY:
The study will include 20 subjects who will be randomly divided to two groups: a ten person group being the study group and a ten person group acting as a control group (each group will include a similar number of females and males as the other group). In addition, the physiotherapy treatments at the rehabilitation center, the study group will gain an intervention consisting of 12 therapy sessions, administered for 12 consecutive days (apart of weekends). The intervention will include 6 minutes of watching a movie clip alternately showing a healthy man and a healthy woman at their sixties, walking while being filmed from various angles. Immediately after watching, the subject will perform 6 minutes of walking, under the experimenters supervision, but without his or hers intervention. Immediately following the walking, the whole procedure will be repeated (watching a clip and walking).

The control group will undergo 12 treatments of the same nature, but will watch the movie clip shown backwards, so that the people filmed will seem to walk backwards (it was established that watching a reversed action does not activate the MNS system activated by a regular execution of the activity [Celnik et al., 2008]), followed by 6 minutes of walking under the experimenters supervision, then watching the movie again and walking again.

The person performing the examinations will be blinded as to the division of the subjects to the study group and the control group. After performing the previously noted examinations needed to participate in the research, the subjects found fit will be examined before the beginning of the intervention, at its end and then three months after its conclusion. The examinations will include smart step and walking parameters.

ELIGIBILITY:
Inclusion Criteria:

* People after a first ischemic or hemorrhagic stroke, up to 60 days following the event.
* A FAC (Functional Ambulation Category) score test result of 2 or 3, in order to ensure basic mobility, even if still requiring supervision.
* A NIHSS (National Institutes of Health Stroke Scale) score of 3 to 18.
* Patients suffering from the following will not be part of the study:

  * Significant neglect (a BIT score under 129 in the conventional tests).
  * Hemianopsy as determined upon a clinical examination by a rehabilitation physician.
  * Clarity of vision problem, determined upon an SC based examination.
  * Significant cognitive decline (a Mini mental test score of under 24).
  * Aphasia which prevents understanding the signing a Helsinki form.

Exclusion Criteria:

* Patients participating in concurrent researches will not participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Smart step examination- Average weight on the hind foot and fore foot. Cycle - time (in seconds) from one initial contact to the other (on the same foot). Stance and swing average percentage of one walking cycle, Cadence | before the beginning of the intervention, at its end and then three months after its conclusion.

SECONDARY OUTCOMES:
2. Two min. walking test. 3. Ten meter walking test. 4. An ABC questioner to determine the personal confidence in regards to walking. | before the beginning of the intervention, at its end and then three months after its conclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Zeev meiner, M.D, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel